CLINICAL TRIAL: NCT06464003
Title: Orthodontic Screening and Treatment Need in Public Health Care
Brief Title: Orthodontic Screening in Public Healthcare
Status: Recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Heidi Arponen, Consultant orthodontist, University of Helsinki
Other Study IDs: UHelsinki
Record Dates: First submitted 2024-06-06; First posted 2024-06-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Malocclusion; Compliance, Patient
MeSH Terms: conditions — Malocclusion; Patient Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Treatment need: Individuals with objective treatment need
  Interventions: Other: Questionnaire
- No treatment need: Individuals with no objectively determined treatment need
  Interventions: Other: Questionnaire
- Controls: Random sample of individuals
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Malocclusion impact questionnaire

SUMMARY:
The aim of the study is to examine orthodontic screening practises in public health care.

DETAILED DESCRIPTION:
The study aims to assess repeatability of malocclusion evaluation in orthodontic treatment need screening in a publicly funded clinic. The objective treatment need is compared with subjective need for orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* residence in the wellbeing services county catchment area
* willingness to participate in the study

Exclusion Criteria:

* Age under 6 years or over 16 years
* insufficient language skills to be able to understand the questionnaire

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Unselected population sample study
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
Treatment need | Baseline
  Orthodontic treatment need

SECONDARY OUTCOMES:
Subjective evaluation | Baseline
  A questionnaire enquiring subjective evaluation of the treatment need and impact of malocclusion on oral heath related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Arponen, Study Director — University of Helsinki
Locations (2):
- Finland (2):
  - University of Helsinki, Helsinki, Helsinki
  - Vantaa and Kerava wellbeing services county, Vantaa, Vantaa

IPD SHARING:
Plan to Share IPD: No